CLINICAL TRIAL: NCT02937545
Title: Delivery of Pharmacogenetic Testing in a Community Pharmacy Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00068552; 2R01GM081416-08A1 (NIH)
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Results first posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Pharmacogenetics
MeSH Terms: interventions — Medication Therapy Management; myotubularin; Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGx Only (Experimental): Patients will receive pharmacogenetic testing. Pharmacists will make recommendations for drug/dose changes based on PGx results.
  Interventions: Other: Pharmacogenetic testing
- PGx + MTM (Experimental): Patients will receive pharmacogenetic testing along with medication therapy management. Two MTM sessions will be conducted: one at the time testing is ordered and the testing sample is collected, and one when results are returned to the patient. Pharmacists will make recommendations for drug/dose changes based on medication action plan developed during MTM and the PGx results.
  Interventions: Other: Medication Therapy Management; Other: Pharmacogenetic testing

INTERVENTIONS:
Other: Medication Therapy Management — Community pharmacists will provide medication therapy management in combination with pharmacogenetic testing
  Other Names: MTM + PGx
  Arms: PGx + MTM
Other: Pharmacogenetic testing — Community pharmacist will provide pharmacogenetic testing.
  Other Names: PGx

SUMMARY:
This study aims to compare patient use of and satisfaction with community pharmacist-delivered pharmacogenetic (PGx) testing delivered along or as part of a medication therapy management (MTM) service. Pharmacist and patient outcome measures will be collected by surveys, interviews, and review of pharmacy records.

DETAILED DESCRIPTION:
This study aims to investigate the delivery of pharmacogenetic (PGx) testing alone or in combination with Medication Therapy Management (MTM) in the community pharmacy setting in order to assess and compare the two delivery models. Using a clust randomized trial, these effects of these two models will be compared. Pharmacist and patient outcome measures will be collected by survey, interviews, and review of pharmacy records. The investigators intend to compare the effect of PGx alone and PGx with MTM from the pharmacy perspective (to assess impact on workflow/operations) and patient perspective (to assess acceptance of testing, understanding of results, medication adherence, and overall satisfaction with delivery model). In the PGx only arm, pharmacists will offer PGx testing to patients who are prescribed one of the 10 eligible drugs (aripiprazole, carisoprodol, celecoxib, citalopram, clopidogrel, metoprolol, nortriptyline, paroxetine, simvastatin, warfarin) and will return results to the patient and physician with any recommendations for drug or dosage changes based on results. In the PGx and MTM arm, pharmacists will offer PGx testing to patients prescribed one of the 10 eligible drugs and provide two MTM sessions: one at the time of testing, and one when results are returned. All patients will be surveyed before PGx testing and 3 months after receiving results. Pharmacists will be surveyed prior to their participation and following the conclusion of the study. Pharmacists will also conduct a chart review of patients and document all interactions with enrolled patients and their providers.

ELIGIBILITY:
Inclusion Criteria:

* Pharmacist participants must be community pharmacists licensed and practicing in North Carolina
* Patient participants must be prescribed one of the 10 eligible medications (aripiprazole, carisoprodol, celecoxib, citalopram, clopidogrel, metoprolol, nortriptyline, paroxetine, simvastatin, warfarin)
* Patient participants must be able to consent to participating and testing on their own, and be able to read English

Exclusion Criteria:

* Patients who have previously undergone pharmacogenetic testing will not be eligible.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled 154 patient participants and 36 pharmacist participants for a total of 190. Patients and pharmacists were assigned to the PGx only or PGx + MTM study arm.
Groups:
- PGx Only (Patients); PGx Only (Pharmacists): Patients received pharmacogenetic testing only. Participating pharmacist made recommendations for drug/dose changes based on PGx results. Data collected from both patients and pharmacists.
- PGx + MTM (Patients): Patients received pharmacogenetic testing along with medication therapy management (MTM). Two MTM sessions will be conducted: one at the time testing is ordered and the testing sample is collected, and one when results are returned to the patient. Pharmacists made recommendations for drug/dose changes based on medication action plan developed during MTM and the PGx results. Data collected from both patients and pharmacists.
  Medication Therapy Management: Community pharmacists will provide medication therapy management in combination with pharmacogenetic testing
- PGx + MTM (Pharmacists): Patients received pharmacogenetic testing plus medication therapy management (MTM). Participating pharmacist made recommendations for drug/dose changes based on PGx results and conducted MTM. Data collected from both patients and pharmacists.
Period: Overall Study
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients) | PGx Only (Pharmacists) | PGx + MTM (Pharmacists)
Started | 69 | 85 | 15 | 21
Completed | 67 | 83 | 9 | 14
Not Completed | 2 | 2 | 6 | 7
Not completed — Withdrawal by Subject | 1 | 2 | 6 | 7
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participating patients who completed the study. No baseline data collected for participating pharmacists.
Groups:
- PGx Only (Patients): Patients will receive pharmacogenetic testing. Pharmacists will make recommendations for drug/dose changes based on PGx results.
  Pharmacogenetic testing: Community pharmacist will provide pharmacogenetic testing.
- PGx + MTM (Patients): Patients will receive pharmacogenetic testing along with medication therapy management. Two MTM sessions will be conducted: one at the time testing is ordered and the testing sample is collected, and one when results are returned to the patient. Pharmacists will make recommendations for drug/dose changes based on medication action plan developed during MTM and the PGx results.
  Medication Therapy Management: Community pharmacists will provide medication therapy management in combination with pharmacogenetic testing
  Pharmacogenetic testing: Community pharmacist will provide pharmacogenetic testing.
- Total: Total of all reporting groups
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients) | Total
Number analyzed (Participants) | 67 | 83 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 38 | 83
  >=65 years | 22 | 45 | 67
Age, Continuous [Mean (Full Range); unit: years] | 57.3 [20 to 84] | 64.2 [23 to 91] | 61.1 [20 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 55 | 89
  Male | 33 | 28 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 7 | 9
  White | 61 | 74 | 135
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 83 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Patient Participants' Acceptance of PGx Services Offered in Community Pharmacy Setting
Description: Post-Study Survey question: "Now that you know your test results, would you have taken the test in the first place?" (Response: 'would definitely' have taken the test)
Time Frame: Post-study Survey (after test results received)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Groups:
- PGx Only (Patients): Received pharmagenetic (PGx) testing from the pharmacist and no additional services (related to the study).
- PGx + MTM (Patients): Received pharmacogenetic (PGx) testing plus medication therapy management (MTM)
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 14 | 13

2. Primary Outcome: Number of Patient Participants Who Recalled All Test Results
Description: Post-Study Survey Question: "As best you can, please choose the result of your drug response test for the following genes" (Response: Result selected for all 5 genes)
Time Frame: Post-study (after test results received)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 13 | 15

3. Primary Outcome: Number of Patient Participants Who Considered Time With Pharmacist to be Worthwhile
Description: Patient survey question - "Did you feel your time spent with the pharmacist was worthwhile?". Reported as number of participants who selected answer choice "Yes, definitely".
Time Frame: Post-study (after test results received)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 16 | 16

4. Primary Outcome: Number of Patient Participants' With High Medication Adherence
Description: Pre-study (baseline) survey question: "In the last 7 days, I took all doses as prescribed" (Response: "strongly agree")
Time Frame: Baseline (prior to testing)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 15 | 12

5. Primary Outcome: Number of Patient Participants With High Medication Adherence (Post-study)
Description: Post-study (follow-up) survey question: "In the last 7 days, I took all doses as prescribed" (Response: "strongly agree")
Time Frame: Post-Study (after test results received)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 11 | 9

6. Primary Outcome: Number of Patient Participants Who Reported Understanding of Implications of Test Results
Description: Post_Study Survey Question: Please indicate your level of agreement with the following statement: "I understood clearly my choices for prevention or early detection of side effects." (Response: "Sometimes/Often")
Time Frame: Post-study (after test results received)
Population: Participants who completed the pre/post-study surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients)
Number analyzed (Participants) | 21 | 17
Participants | 11 | 16

7. Secondary Outcome: Number of Pharmacist Participants Who Reported Strong Likelihood to Continue to Deliver PGx Testing
Description: Pharmacist Post-Survey Question: How likely are you to continue providing PGx testing in your pharmacy after the conclusion of the study? (Answer response: "definitely continue")
Time Frame: Post-study (3 months)
Population: Pharmacists who completed the survey.
Measure: Count of Participants; unit: Participants
Groups:
- PGx Only (Pharmacists): Pharmacists delivered PGx only tests to eligible/consented patients
- PGx + MTM (Pharmacists): Pharmacists delivered PGx testing with MTM to eligible/consented patients
Arm/Group | PGx Only (Pharmacists) | PGx + MTM (Pharmacists)
Number analyzed (Participants) | 7 | 9
Participants | 0 | 2

8. Secondary Outcome: Average Score of PGx Knowledge Assessment by Pharmacist Participants
Description: 7-question knowledge assessment of pharmacogenetics. Possible Score Range 0-7; actual range 3-7 (higher scores correspond to higher number of correct answers/higher knowledge)
Time Frame: Baseline (prior to start of study)
Population: All participating pharmacists.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- PGx Plus MTM (Pharmacists): Pharmacists delivered PGx testing with MTM to eligible/consented patients
Arm/Group | PGx Only (Pharmacists) | PGx Plus MTM (Pharmacists)
Number analyzed (Participants) | 15 | 21
score on a scale | 5.4 [4 to 7] | 5.3 [3 to 7]

9. Secondary Outcome: Number of Pharmacist Participants Who Reported 'Reimbursement' as Most Common Barrier to Delivery of PGx Testing
Description: Pharmacist Post-Survey Question: Of the following potential barriers to providing PGx testing services, please indicate the greatest perceived barrier (most common response: "reimbursement")
Time Frame: Post-study (3 months)
Population: Pharmacists who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Pharmacists) | PGx + MTM (Pharmacists)
Number analyzed (Participants) | 7 | 9
Participants | 5 | 3

10. Secondary Outcome: Number of Participating Pharmacists Who Feel Qualified to Deliver PGx Testing
Description: Pharmacist Post-Study survey question: I feel qualified to provide PGx testing at my pharmacy (Answer response: "strongly agree/agree").
Time Frame: Post-study (3 months)
Population: Pharmacists who completed the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | PGx Only (Pharmacists) | PGx + MTM (Pharmacists)
Number analyzed (Participants) | 7 | 9
Participants | 7 | 7

ADVERSE EVENTS:
Time Frame: Data collected from enrollment through 6 months follow-up.
Groups:
- PGx Only (Pharmacists): Participating pharmacists provided participating patients with pharmacogenetic testing only
- PGx + MTM (Pharmacists): Participating pharmacists provided participating patients with pharmacogenetic testing along with medication therapy management (MTM)
Arm/Group | PGx Only (Patients) | PGx + MTM (Patients) | PGx Only (Pharmacists) | PGx + MTM (Pharmacists)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/83 | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/83 | 0/15 | 0/21
Other Adverse Events (participants affected / at risk) | 0/67 | 0/83 | 0/15 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT02937545/Prot_SAP_000.pdf